CLINICAL TRIAL: NCT06638580
Title: Periodontitis Provokes Retinal Neurodegenerative Effects of Metabolic Syndrome: A Cross-Sectional Study
Status: Completed | Type: Observational
Sponsor: Recep Tayyip Erdogan University (Other)
Responsible Party: Principal Investigator, Hatice Yemenoglu, Assistant Professor, Recep Tayyip Erdogan University
Other Study IDs: 2022/157
Record Dates: First submitted 2024-10-08; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Periodontitis; Metabolic Syndrome; Neurodegeneration; Oxidative Stress; Optic Coherence Tomography
Keywords: periodontitis; metabolic syndrome; neurodegeneration; oxidative stress; optic coherence tomography
MeSH Terms: conditions — Periodontitis; Metabolic Syndrome; Nerve Degeneration

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples Without DNA — serum
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Control: Systemically and periodontally healthy
  Interventions: Diagnostic Test: Clinical Periodontal Measurements (plaque index, gingival index, bleeding index, clinical attachment level), Optical Coherence Tomographic Measurements, Serum IL1-β, TNF-α, IL-10, TAS, TOS, OSİ levels
- PD: systemically healthy periodontitis
  Interventions: Diagnostic Test: Clinical Periodontal Measurements (plaque index, gingival index, bleeding index, clinical attachment level), Optical Coherence Tomographic Measurements, Serum IL1-β, TNF-α, IL-10, TAS, TOS, OSİ levels
- MetS: periodontally healthy metabolic syndrome
  Interventions: Diagnostic Test: Clinical Periodontal Measurements (plaque index, gingival index, bleeding index, clinical attachment level), Optical Coherence Tomographic Measurements, Serum IL1-β, TNF-α, IL-10, TAS, TOS, OSİ levels
- PD-MetS: periodontitis and metabolic syndrome combined
  Interventions: Diagnostic Test: Clinical Periodontal Measurements (plaque index, gingival index, bleeding index, clinical attachment level), Optical Coherence Tomographic Measurements, Serum IL1-β, TNF-α, IL-10, TAS, TOS, OSİ levels

INTERVENTIONS:
Diagnostic Test: Clinical Periodontal Measurements (plaque index, gingival index, bleeding index, clinical attachment level), Optical Coherence Tomographic Measurements, Serum IL1-β, TNF-α, IL-10, TAS, TOS, OSİ levels — Probing pocket depth (PPD) was measured as the distance between the deepest point of the sulcus (or pocket) and the gingival margin, and clinical attachment level (CAL) was measured as the distance between the base of the pocket and the cementoenamel junction. PPD and CAL were measured at six different points (mesio-buccal, mid-buccal, disto-buccal, mesio-lingual, mid-lingual, and disto-lingual) in each tooth, and other index scores were taken at four different points (mesial, distal, vestibular and palatinal).
  Serum IL1-β, TNF-α, and IL-10 levels were measured via immunosorbent assay method using human-specific kits according to the kit manufacturer's instructions.
  Serum total antioxidant status (TAS) and total oxidant status (TOS) levels were mea-sured by a spectrophotometric method using specific kits.
  Retinal and choroidal imaging and measurements were performed with optical coherence tomography (SS-OCT) with swept-source (SS) technology and non-invasive OCT angiography.

SUMMARY:
This cross-sectional study aimed to investigate the retino-choroidal degenerative effects of periodontitis, metabolic syndrome (Mets), and the combination of these diseases using optical coherence tomography (OCT) measurements. Methods: Ninety-two patients selected according to inclusion criteria were divided into 4 groups: systemically and periodontally healthy (Control), systemically healthy periodontitis (PD), periodontally healthy metabolic syndrome (MetS), and periodontitis and metabolic syndrome combined (PD-MetS). The systemic inflammatory-oxidative effects of periodontitis and MetS were biochemically evaluated using serum TNF (Tumor necrosis factor)-α level, IL(Interleukin)-1β/IL-10 ratio, and oxidative stress index (OSI: TOS/TAS). Retinal (AMT, peripapillary retinal nerve fiber layer thickness (pRNFLT), and Ganglion cell and Inner plexiform layers (GCL+T) and choroidal (SFCT) morphometric measurements and vascular evaluations (foveal capillary density) were performed via OCT Angio with swept-source technology.

To the best of our knowledge, although there are many clinical studies on the possible effects of Mets on retino-choroidal layers, there is a limited amount of evidence on the effects of periodontitis which is from an animal study. Moreover, there are no studies on the retinal degenerative effects of the combined presence of periodontitis and Mets. In this context, the present study is unique and based on the hypothesis that the alone or combined presence of periodontitis and Mets may provoke retino-choroidal degenerative changes through systemic inflammatory stress.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with stage III/IV, grade C periodontitis,
* Patients with at least 20 teeth,
* Patients diagnosed with MetS,
* Obese [waist circumference (WC) 80 cm ≥ for women and 94 cm ≥ for men], Type 2 (Diabetes Mellitus) DM and hypertensive patients.

Exclusion Criteria:

* Cancer,
* Any autoimmune disease,
* Osteoporosis,
* Active infectious disease (acute hepatitis, tuberculosis, AIDS),
* Vitreoretinal, optic nerve or choroidal vascular disease,
* Acute and chronic ocular diseases (such as cataract, glaucoma, macular degeneration, uveitis, Behçet's, scleritis),
* History of refractive or intraocular surgery,
* Immunosuppressive, oral contraceptive, bisphosphonate and antioxidant drug use,
* Pregnancylactation,
* Smokers.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Rize, Türkiye
Sampling Method: Non-Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-10-30 (Actual)

PRIMARY OUTCOMES:
optical coherence tomography (OCT) | 6 months
  Retinal and choroidal imaging and measurements will perform with it.

SECONDARY OUTCOMES:
probing pocket depth (PPD) | 6 months
  It measures as the distance between the deepest point of the sulcus (or pocket) and the gingival margin
clinical attachment level (CAL) | 6 months
  CAL will measure as the distance between the base of the pocket and the cemento-enamel junction.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Ophthalmology of the Faculty of Medicine of Recep Tayyip Erdogan University, Rize, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual data may be shared if requested with reasonable justification.